CLINICAL TRIAL: NCT07000760
Title: Intraoperative Ultrasonic Atomization of Lidocaine and Postoperative Pulmonary Complications
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jun Zhang (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2504-Exp179
Record Dates: First submitted 2025-05-22; First posted 2025-06-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pulmonary Complications (PPCs)
Keywords: Postoperative pulmonary complications; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine (Experimental): After anesthetic induction and before the end of the surgery, 100mg of 2% lidocaine was nebulized and inhaled respectively.
  Interventions: Drug: Ultrasonic atomization of lidocaine
- saline (Placebo Comparator): After anesthetic induction and before the end of the surgery, the same volume of normal saline (5ml of 0.9% NaCl) was ultrasonically atomized.
  Interventions: Drug: Ultrasonic atomization of normal saline

INTERVENTIONS:
Drug: Ultrasonic atomization of lidocaine — After induction of general anesthesia and before the end of the surgery, 100mg of 2% lidocaine was nebulized and inhaled respectively, and the nebulization time was 15-20 minutes each time.
  Other Names: 1
  Arms: lidocaine
Drug: Ultrasonic atomization of normal saline — After anesthesia induction and before the end of the surgery, the same volume of normal saline (5ml of 0.9% NaCl) was ultrasonically atomized, and the atomization time was 15-20 minutes each time.
  Other Names: 2
  Arms: saline

SUMMARY:
There is high incidence of postoperative pulmonary complications (PPCs) in patients undergoing major abdominal surgeries.PPCs significantly prolongs the hospital stay of patients, increases their economic burden, and raises the mortality rates within 30 days and 1 year after surgery. The inflammatory response during the perioperative period plays an important role in the occurrence and development of PPCs. The anti-inflammatory effect of lidocaine has a potential lung protection mechanism. The purpose of this study is to explore the effect of ultrasonic atomization of lidocaine on the incidence of PPCs. The investigators hypothesized that intraoperative ultrasonic atomization of lidocaine could reduce the incidence of PPCs.

DETAILED DESCRIPTION:
Introduction Globally, over 313 million surgical procedures are performed annually, with postoperative pulmonary complications (PPCs) occurring in 5-33% of cases. PPCs, the second most common postoperative complication after surgical site infections, encompass conditions such as respiratory infections, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, and aspiration pneumonia. These complications significantly prolong hospital stays, increase healthcare costs, and elevate 30-day and 1-year mortality rates.

Pathophysiology of PPCs PPCs are closely linked to perioperative pulmonary inflammatory responses. Mechanical ventilation during general anesthesia alters pulmonary ventilation distribution, leading to atelectasis in over 90% of patients. Atelectasis increases mechanical stress and hypoxia in collapsed lung regions while causing hyperinflation and hyperoxia in adjacent areas. These conditions promote the release of pro-inflammatory cytokines, reactive oxygen species, and leukocyte infiltration. Additionally, atelectasis-induced hypoxia and mechanical stress contribute to endothelial damage, increasing vascular permeability and protein leakage. Major abdominal and thoracic surgeries further exacerbate systemic inflammation and airway hyperreactivity, impairing alveolar epithelial barrier function and mucociliary clearance.

Lidocaine's Anti-Inflammatory and Lung-Protective Mechanisms Lidocaine has emerged as a potential therapeutic agent due to its anti-inflammatory properties. Studies indicate that it inhibits neutrophil infiltration and reduces pro-inflammatory cytokines (e.g., IL-6, TNF-α) by blocking Toll-like receptor 4/NF-κB signaling. Inhaled lidocaine has shown efficacy in murine asthma models by suppressing GATA-3 expression, eosinophilic inflammation, mucus overproduction, and airway hyperreactivity. It has also been explored as an adjunct therapy for severe COVID-19 respiratory symptoms, mitigating cytokine storms and improving outcomes. In pediatric patients, lidocaine reduces postoperative cough incidence.

Current Challenges and the Promise of Ultrasonic Nebulization Despite its potential, lidocaine's clinical application for lung protection remains inconsistent. Intravenous administration poses risks due to narrow therapeutic windows, with fluctuating plasma concentrations potentially causing neurotoxicity or cardiotoxicity. Conventional nebulizers produce particles >5 μm, depositing primarily in the upper airways, with less than 15% reaching the lung parenchyma. In contrast, ultrasonic nebulization generates 1-5 μm aerosol particles, enhancing lower respiratory tract deposition to 40-60%. Animal studies demonstrate that nebulized lidocaine achieves lung tissue concentrations 8-10 times higher than plasma levels, suggesting targeted efficacy.

Research Objective and Hypothesis The role of ultrasonic nebulized lidocaine in reducing PPCs remains underexplored. This study aims to evaluate its impact on PPC incidence within seven days post-surgery. The hypothesis is that intraoperative ultrasonic nebulized lidocaine administration will decrease PPC rates, offering a safer and more effective approach to perioperative lung protection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed the informed consent form and are willing to complete the study according to the protocol
* Age ≥18 years old and ≤90 years old
* ASA classification grades I-III
* Elective major non-cardiac surgery
* General anesthesia under tracheal intubation
* Monitor invasive arterial blood pressure
* The expected operation time ≥2 hours

Exclusion Criteria:

* Untreated ischemic heart disease Severe cardiovascular and cerebrovascular diseases
* Severe asthma, pulmonary bullae, pneumothorax, bronchopleural fistula, etc
* Severe underlying liver and kidney diseases
* Age under 18 years old or over 90 years old
* The expected operation time is ≥2 hours

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2025-12-06 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of PPCs within seven days after surgery | Up to one week

SECONDARY OUTCOMES:
ICU admission rate | Up to one week
Hospital stay | Perioperative
Postoperative pain score | Up to one week
  Postoperative pain was assessed using the Visual Analog Scale (VAS), where 0 indicates no pain and 10 represents the most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang Fudan University Shanghai Cancer Centre, Professor, Study Chair — Fudan University Shanghai Cancer Centre
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Centre, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai

IPD SHARING:
Plan to Share IPD: No
The data sets are available from the corresponding author on reasonable request.